CLINICAL TRIAL: NCT02893579
Title: Smartphone-delivered Stress Reduction Intervention for Women With Ischemic Heart Disease
Brief Title: Stress Reduction Intervention for Women With Ischemic Heart Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: were not able to find enough eligible patients. We recruited 6, with incomplete data on those participants.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-00650
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (Experimental): Stress reduction intervention 1 time a month
  Interventions: Behavioral: Early SR intervention
- Delayed Intervention (Experimental): Wait list Control
  Interventions: Behavioral: Delayed SR intervention

INTERVENTIONS:
Behavioral: Early SR intervention — Self-directed stress reduction program delivered through a smart-phone application
  Arms: Early Intervention
Behavioral: Delayed SR intervention — Activity tracking only for the first month
  Arms: Delayed Intervention

SUMMARY:
This is a single center, randomized controlled trial which will include women with ischemic heart disease to receive either a self-directed stress reduction program delivered through a smart-phone application or activity tracking only for the first month ("early SR intervention" and "delayed SR intervention", respectively). Patients will be monitored for 1 month for application use and step counts via telephone or email interview and/or collection of screen-captured data. Baseline questionnaires will be repeated at the end of one month to assess for all primary and secondary measures, at which time the control group (activity tracking only) will be introduced to the intervention program. The early SR intervention group will not receive a new intervention but will be encouraged to continue using the app. Data will be collected for an additional 2 months with all participants in both groups. After the three-month study period, the study will close with the collection of final questionnaire data.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ischemic heart disease as defined by one or more of the following within the last 2 years:
* Positive stress test
* Admission for ACS, PCI, or CABG
* Typical or atypical ischemic symptoms within one month of enrollment
* On stable dose of anti-anginal medications for at least 2 months
* Able and willing to provide informed consent and comply with all aspects of the protocol
* Owns a smartphone with the ability to download applications for stress reduction and activity tracking
* English-speaking (apps are not available in other languages)

Exclusion Criteria:

* Planned for revascularization during the study period
* Self-reported or chart-reviewed diagnosis of psychotic disorder including schizophrenia or schizoaffective disorder, bipolar disorder
* Current participation in a cardiac rehab program or planned participation during the study period

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire [SAQ] | Change from Baseline to 3 Months
  The Seattle Angina Questionnaire is a well-validated descriptive instrument for measuring quality of life across five dimensions of coronary artery disease: physical limitation, anginal stability, anginal frequency, treatment satisfaction and disease perception. 45 Patient SAQ scores have been found to be independently prognostic of subsequent mortality, hospitalization, and resource use.
Rose Dyspnea Score | Change from Baseline to 3 Months
  The Rose Dyspnea Score provides additional information about patient dyspnea, which is a common complaint in patients with IHD independent of the presence of heart failure.
Patient Health Questionnaire [PHQ-2] | Change from Baseline to 3 Months
  a 2-item screening tool for depression, which can be assessed further using the Patient Health Questionnaire-9 if positive

SECONDARY OUTCOMES:
Duke Activity Status Index score | Change from Baseline to 3 Months
  independently and incrementally predicts major adverse cardiac events (MACE) in patients post-MI as well as in those with chronic stable heart failure
European Quality of Life- Five Dimensions (EQ-5D) scores | Change from Baseline to 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States